CLINICAL TRIAL: NCT00466505
Title: A Phase 2 Study of Cetuximab in Combination With Celecoxib in Colorectal Cancer
Brief Title: Cetuximab & Celecoxib for Metastatic Colorectal Cancer or Colorectal Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jordan Berlin, MD, Jordan Berlin, MD, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0410; P30CA068485 (NIH); VU-VICC-GI-0410; VU-IRB-040227
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2011-11-16 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Celecoxib; Immunohistochemistry; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental)
  Interventions: Biological: cetuximab; Drug: celecoxib; Genetic: proteomic profiling; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: mass spectrometry

INTERVENTIONS:
Biological: cetuximab — 400 mg/m2 iv week 1, then 250 mg/m2 weekly thereafter, starting on day 1 and continuing until progressive disease, excessive toxicity or removal from study for other reasons listed in the protocol.
  Other Names: Erbitux, IMC-C225
Drug: celecoxib — 200 mg po BID starting on day 1 and continuing until progressive disease, excessive toxicity or removal from study for other reasons listed in the protocol.
  Other Names: celebrex
Genetic: proteomic profiling — Serum samples obtained as above will be analyzed by proteomic analysis in order to determine biomarkers of treatment response and toxicity prediction. We will use LC-MS-MS or MALDITOF mass spectrometry.
Other: immunohistochemistry staining method — phospho-EGFR levels using western blots of tissue extracts and immunohistochemistry on frozen and (if no other option available, paraffinembedded tissue sections).
Other: laboratory biomarker analysis — Serum samples obtained as above will be analyzed by proteomic analysis in order to determine biomarkers of treatment response and toxicity prediction.
Other: mass spectrometry — We will use LC-MS-MS or MALDITOF mass spectrometry. Before any tissues are received, the drug of interest is evaluated via MALDI mass spectrometry on a MDS/Sciex QStar QqTOF mass spectrometer.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving cetuximab together with celecoxib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with celecoxib works in treating patients with metastatic colorectal cancer or colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in patients with unresectable or metastatic colorectal cancer treated with cetuximab and celecoxib.

Secondary

* Determine the response rate, median survival, and 1-year survival rate of patients treated with this regimen.
* Determine the toxicity profile of this regimen in these patients.
* Determine the feasibility of testing urinary PGE-M in patients treated with this regimen.
* Determine the feasibility of testing serum transforming growth factor-α and amphiregulin in patients treated with this regimen.
* Determine the effects of this regimen on the EGFR pathway in tumor cells (i.e., phosphorylated EGFr, phosphorylated AKT, activated mitogen-activated protein kinase).
* Determine the effects of this regimen on the cyclooxygenase-2 pathway in tumor cells by measuring PGE-2 levels.

OUTLINE: Patients receive cetuximab IV over 1-2 hours once weekly and oral celecoxib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Serum and urine samples are collected at baseline, after week 1, and every other course thereafter for evaluation of PGE-2 by mass spectrometry, cyclooxygenase-2 activity, and phospho-EGFR levels by western blot analysis and immunohistochemistry. Samples are also analyzed for TGF-α and amphiregulin proteomics.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed colorectal cancer that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > or equal to 20 mm with conventional techniques or as > or equal 10 mm with spiral CT scan.
* Patients must have progressed after at least 1 chemotherapy regimen for advanced disease. No prior therapy which specifically and directly targets the EGFR pathway.
* Age 18 years or older
* ECOG performance status ≤ 2.
* Life expectancy of greater than 3 months.
* Normal organ and marrow functions as defined below:

  * absolute neutrophil count ≤ 1,500/μl
  * platelets ≤ 100,000/μl
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) > or equal to 2.5 times institutional upper limit of normal or > or equal to 5.0 times normal if liver metastases are present
  * creatinine within normal institutional limits OR
  * creatinine clearance > or equal to 60 mL/min/1.73 m2 for patients creatinine levels above institutional normal
* The effects of cetuximab and/or celecoxib on the developing human fetus at the recommended therapeutic doses are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to provide written informed consent.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Prior severe infusion reaction to a monoclonal antibody
* Serum calcium >12.0 mg/dl.
* Patients must be off all other selective or non-selective COX-2 inhibitors for at least 2 weeks prior to study entry (with the exception of 81 mg of daily aspirin).
* No major surgery within 4 weeks. No minor surgery (laparoscopy, thoracoscopy, port placement) within 1 week.
* Patients must be > 4 weeks from prior pelvic radiation and recovered from side effects.
* Patients must be > 1 week from prior palliative radiation and have recovered from all side effects.
* Prior treatment with EGFR targeting therapies.
* Significant traumatic injury occurring within 28 days prior to treatment.
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because cetuximab is an epidermal growth factor inhibitor with the potential for teratogenic or abortifacient effects based on the data suggesting that EGFR expression is important for normal organ development. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cetuximab, breastfeeding should be discontinued if the mother is treated with cetuximab.
* Patients with known HIV disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-05; Primary Completion 2008-07 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan D. Berlin, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment period was May 2005 through January 2007.
Pre-assignment Details: A total of 18 people signed consent to participate in this study. One was determined ineligible, for a total of 17 patients on study.
Period: Overall Study
Arm/Group | Therapeutic Intervention
Started | 17
Completed | 0
Not Completed | 17
Not completed — disease progression | 13
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Number of days from study enrollment to evidence of progressive disease radiographically, with progression defined under RECIST criteria as at least 20% increase in sum of longest diameter of target lesions
Time Frame: On study date to off study date in this study with median 9.76 months
Measure: Median (Full Range); unit: Days
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 17
Days | 55 [10 to 295]

2. Secondary Outcome: Patient Response to Treatment
Description: Number of patients in each response category according to RECIST criteria: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: On study date to off study date in this study with median 9.76 months
Measure: Number; unit: participants
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 17
participants
  Partial Response | 2
  Progressive Disease | 7
  Stable Disease | 4
  Unknown | 4

3. Secondary Outcome: Overall Survival
Description: Median survival time in months, from on-study date to date of death
Time Frame: On study date to off study date in this study with median 9.76 months
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 17
Months | 8.54 [5.58 to 10.74]

4. Secondary Outcome: One Year Survival Rate
Description: Percent of patients who remain alive one year from on-study date
Time Frame: 1 year from on-study date
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 17
Percentage of participants | 17.6 [6.32 to 49.3]

5. Secondary Outcome: Number of Patients With Each Worst-grade Toxicity Response
Description: Number of patients with worst-grade toxicity response of each grade (grade 1 to 5) following NCI Common Toxicity Criteria, with grade 1=mild adverse event; 2=moderate adverse event; 3=severe and undesirable adverse event; 4=life-threatening or disabling adverse event; 5=death.
Time Frame: On study date to off study date in this study with median 9.76 months
Measure: Number; unit: patients
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 17
patients
  No. of patients with worst-grade toxicity of 1 | 0
  No. of patients with worst-grade toxicity of 2 | 0
  No. of patients with worst-grade toxicity of 3 | 1
  No. of patients with worst-grade toxicity of 4 | 1
  No. of patients with worst-grade toxicity of 5 | 0

6. Secondary Outcome: Urinary PGE-M : Treatment Cycle 1
Description: Measurement in ng/mL of a stable metabolite of prostaglandin E2 (PGE-M) in urine during treatment cycle 1
Time Frame: on-study week 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 17
ng/mL
  Stable or PR (n=6) | 30.42 (17.15)
  Progressive Disease (n=11) | 21.94 (17.13)

7. Secondary Outcome: Serum TGF-alpha: Treatment Cycle 1
Description: Measurement in ng/mL of tumor growth factor-alpha (TGF-alpha) in serum samples during treatment cycle 1
Time Frame: on-study week 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 17
ng/mL
  Stable or PR (n=5) | 26.38 (17.15)
  Progressive Disease (n=10) | 25.90 (10.93)

8. Secondary Outcome: Urinary PGE-M : Treatment Cycle 2
Description: Measurement in ng/mL of a stable metabolite of prostaglandin E2 (PGE-M) in urine during treatment cycle 2
Time Frame: on-study week 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 17
ng/mL
  Stable or PR (n=6) | 28.42 (25.73)
  Progressive Disease (n=4) | 29.76 (41.34)

9. Secondary Outcome: Serum TGF-alpha: Treatment Cycle 2
Description: Measurement in ng/mL of tumor growth factor-alpha (TGF-alpha) in serum samples during treatment cycle 2
Time Frame: on-study week 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 17
ng/mL
  Stable or PR (n=6) | 48.02 (16.94)
  Progressive Disease (n=4) | 49.95 (27.27)

ADVERSE EVENTS:
Arm/Group | Therapeutic Intervention
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Intervention (N=17)
Hemorrhage, bladder (Renal and urinary disorders) | 1 (1)
neurology, brain mets (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Intervention (N=17)
hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
alkaline phosphatase (Investigations) | 4 (5)
allergic reaction (General disorders) | 3 (3)
ALT, SGPT (Metabolism and nutrition disorders) | 2 (2)
anorexia (Psychiatric disorders) | 4 (4)
AST, SGOT (Blood and lymphatic system disorders) | 3 (3)
hyperbilirubinemia (Metabolism and nutrition disorders) | 3 (3)
hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
edema (General disorders) | 2 (3)
cataract (Eye disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 4 (4)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
dermatologic general (Skin and subcutaneous tissue disorders) | 7 (8)
diarrhea (Gastrointestinal disorders) | 7 (8)
dizziness (Nervous system disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
fatigue (General disorders) | 12 (13)
dyspepsi (Gastrointestinal disorders) | 3 (3)
hemoglobin (Investigations) | 7 (11)
hemorrhage, rectum (Gastrointestinal disorders) | 3 (3)
hemorrhage, bladder (Renal and urinary disorders) | 4 (4)
hemorrhage, pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hemorrhoids (Gastrointestinal disorders) | 1 (1)
hot flashes (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 (1)
anal incontinence (Gastrointestinal disorders) | 1 (1)
infection (Infections and infestations) | 3 (3)
infection with normal ANC (Infections and infestations) | 1 (1)
insomnia (Psychiatric disorders) | 4 (4)
leukocytes (Blood and lymphatic system disorders) | 1 (1)
hypomagnesiumia (Metabolism and nutrition disorders) | 6 (6)
hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)
agitation (Psychiatric disorders) | 2 (2)
depression (Psychiatric disorders) | 2 (2)
muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
reflux (Gastrointestinal disorders) | 2 (2)
hyperglycemia (Metabolism and nutrition disorders) | 4 (5)
nail changes (Skin and subcutaneous tissue disorders) | 2 (3)
restless leg (Nervous system disorders) | 2 (2)
balanitis (Skin and subcutaneous tissue disorders) | 2 (2)
peripheral neuropathy (Nervous system disorders) | 5 (5)
eye irritation (Eye disorders) | 2 (3)
pain, abdominal (Gastrointestinal disorders) | 8 (8)
pain, back (Musculoskeletal and connective tissue disorders) | 3 (3)
pain, extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
pain, head (Nervous system disorders) | 1 (1)
pain, muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
pain, rib cage (Musculoskeletal and connective tissue disorders) | 2 (2)
pain, rectum (Gastrointestinal disorders) | 2 (2)
platelets (Investigations) | 2 (2)
pruritus, itching (Skin and subcutaneous tissue disorders) | 5 (5)
rash, desquamation (Skin and subcutaneous tissue disorders) | 15 (20)
hand, foot rash (Skin and subcutaneous tissue disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 5 (5)
urinary frequency (Renal and urinary disorders) | 2 (2)
urinary retention (Renal and urinary disorders) | 2 (2)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
diaphoresis, sweating (Vascular disorders) | 2 (2)
tremor (Nervous system disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
vaginal discharge (Reproductive system and breast disorders) | 1 (1)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
blurred vision (Eye disorders) | 2 (2)
flatulence (Gastrointestinal disorders) | 1 (1)
fever (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes